CLINICAL TRIAL: NCT02180438
Title: An Open Label Trial of STRIBILD™ (Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate) for ARV-naïve HIV-2 Infected Adults in Dakar, Senegal
Brief Title: An Open Label Trial of Stribild for Antiretroviral (ARV)-naïve HIV-2 Infected Adults in Dakar, Senegal
Acronym: Stribild HIV-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Clinique des Maladies Infectieuses Ibrahima DIOP Mar/CRCF, Centre Hospitalier Universitaire de Fann (Unknown); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Geoffrey S. Gottlieb, Associate Professor, Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000757
Record Dates: First submitted 2014-05-29; First posted 2014-07-02 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: HIV-2 Infection
Keywords: HIV-2
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; elvitegravir; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open label prospective single arm study of Stribild (Experimental)
  Interventions: Drug: Stribild (Elvitegravir/Cobicistat/Emtricitabine/Tenofovir DF) 1 tablet daily X 48 weeks

INTERVENTIONS:
Drug: Stribild (Elvitegravir/Cobicistat/Emtricitabine/Tenofovir DF) 1 tablet daily X 48 weeks

SUMMARY:
There is a critical need for safe and effective antiretroviral treatment (ART) regimens for HIV-2 infection. This is especially true in West Africa, where the vast majority of the 1-2 million individuals infected with HIV-2 live and were access to effective ART for HIV-2 is limited. HIV-2 is intrinsically resistant to non-nucleoside reverse transcriptase inhibitors (NNRTI) and the fusion inhibitor enfuvirtide (T-20) and mutations conferring broad resistance to nucleoside/nucleotide reverse transcriptase inhibitors (NRTI) are frequently observed in HIV-2 from patients receiving ART. Although antiretroviral protease inhibitors (PI) can be used effectively to treat HIV- 2, HIV-1 and HIV-2 also exhibit important differences in their susceptibilities with studies indicating that saquinavir (SQV), lopinavir (LPV), and darunavir (DRV) are the only potent PI's against HIV-2 replication and cross-resistance is frequent. Although an increasing body of evidence supports the potential utility of integrase inhibitors (INI) against HIV-2, there have been no clinical trials to assess their effectiveness and they are not routinely available in resource-limited settings. These limitations present major challenges to HIV-2 treatment, particularly in the areas in which it is most prevalent. This study is the 1st use of STRIBILD (elvitegravir (EVG), cobicistat (COBI), emtricitabine (FTC), tenofovir disoproxil fumarate (TDF)), an INI-based single tablet regimen, in HIV-2 infected adults in West Africa. The investigators hypothesize STRIBILD will be safe and effective as ART for HIV-2 infection. The Specific Aims of this study are: AIM 1: A pilot, open label, 48 week trial of STRIBILD (elvitegravir, cobicistat, emtricitabine, tenofovir disoproxil fumarate) in 30 ARV-naïve HIV-2 Infected Adults in Dakar, Senegal. AIM 2: Determination of genotypic and phenotypic HIV-2 antiretroviral resistance in individuals with virologic failure (HIV-2 plasma RNA >250 copies/ml) participating in the 48 week trial of STRIBILD

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years old
* HIV-2 Infection (confirmed by DetermineTM & Immunocomb II)
* ARV-naïve
* CD4 count < 750 cells/mm3 and/or WHO Stage 3 or 4 disease
* Anticipate residing in Dakar area for duration of study

Exclusion Criteria:

* Pregnancy or Breast feeding
* HIV-1 or HIV-1/HIV-2 dual infection
* Known allergy or contraindication to Elvitegravir, Cobicistat, Emtricitabine, or Tenofovir DF
* Active Tuberculosis (STRIBILD contraindicated with rifampin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey S Gottlieb, MD PhD, Principal Investigator — University of Washington; Moussa Seydi, MD, Principal Investigator — Clinique des Maladies Infectieuses Ibrahima DIOP Mar/CRCF, Centre Hospitalier Universitaire de Fann
Locations (1):
- Clinique des Maladies Infectieuses Ibrahima DIOP Mar/CRCF, Centre Hospitalier Universitaire de Fann, Dakar, Senegal

REFERENCES:
- [Derived] Ba S, Raugi DN, Smith RA, Sall F, Faye K, Hawes SE, Sow PS, Seydi M, Gottlieb GS; University of Washington-Dakar HIV-2 Study Group. A Trial of a Single-tablet Regimen of Elvitegravir, Cobicistat, Emtricitabine, and Tenofovir Disoproxil Fumarate for the Initial Treatment of Human Immunodeficiency Virus Type 2 Infection in a Resource-limited Setting: 48-Week Results From Senegal, West Africa. Clin Infect Dis. 2018 Oct 30;67(10):1588-1594. doi: 10.1093/cid/ciy324. PMID 29672676

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Prospective Single Arm Study of Stribild: Stribild (Elvitegravir/Cobicistat/Emtricitabine/Tenofovir DF) 1 tablet daily X 48 weeks
Period: Overall Study
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Started | 30
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 49 [24 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Senegal | 30

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: Number of Participants Experiencing Death within the study period
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 0

2. Primary Outcome: New WHO Stage 3 or 4 Event
Description: New AIDS defining event per WHO criteria
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 0

3. Primary Outcome: Virologic Failure, FDA Snapshot (HIV-2 Plasma Viral Load >50 and >400 Copies/ml)
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants
  >50 copies/mL | 1
  >400 copies/mL | 0

4. Secondary Outcome: Grade 3 or 4 Adverse Events
Description: Adverse event per NIH/DAIDS criteria
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants
  Lab: Grade 3 or 4 | 7
  Clinical: Grade 3 or 4 | 1

5. Secondary Outcome: CD4 T-cell Count at 48 Weeks < Baseline
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 0

6. Secondary Outcome: < 50 CD4 T-cell Increase at 48 Weeks From Baseline
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 2

7. Secondary Outcome: Switching Off Stribild Prior to 48 Weeks
Time Frame: 48 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 0

8. Secondary Outcome: Development of Drug Resistance Mutations to Elvitegravir or Emtricitabine or Tenofovir DF
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 1

9. Other Pre Specified Outcome: Interim 24 Weeks Analysis of Death
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
participants | 0

10. Other Pre Specified Outcome: Interim Analysis at 24 Weeks of New WHO Stage 3 or 4 Event
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 0

11. Other Pre Specified Outcome: Interim Analysis at 24 Weeks of HIV-2 Virologic Failure
Description: Virologic failure, FDA Snapshot (HIV-2 plasma viral load >50 and >400 copies/ml)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 0

12. Other Pre Specified Outcome: Interim Analysis at 24 Weeks of Grade 3 and 4 Adverse Events
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Arm/Group | Open Label Prospective Single Arm Study of Stribild
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Prospective Single Arm Study of Stribild (N=30)
CVA (Nervous system disorders) | 1 (1) — stroke

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No